CLINICAL TRIAL: NCT07224529
Title: Efficacy of Vevye Ophthalmic Solution for the Treatment of Meibomian Gland Dysfunction
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Harrow Inc (Industry)
Responsible Party: Principal Investigator, Jillian Ziemanski, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 300015544
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Meibomian Gland Dysfunction (MGD)
Keywords: Dry Eye Disease, Ocular surface inflammation, Tear film Instability; corneal staining; Meibomian Gland Dysfunction; Vevye
MeSH Terms: conditions — Meibomian Gland Dysfunction; Dry Eye Syndromes | interventions — Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a non-randomized, open-label, single-arm interventional study in which all participants receive Vevye® (cyclosporine 0.1%) twice daily in both eyes for 24 weeks following a 2-week artificial-tear run-in period.
Masking Description: All participants, investigators, and study staff will know the treatment being administered. No masking or blinding procedures are implemented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Participants will receive Vevye® (cyclosporine 0.1% ophthalmic solution) twice daily in both eyes for 24 weeks, following a 2-week run-in period using a commercially available artificial tear.
  All participants will undergo standardized ocular assessments including Visual Analog Scale (VAS) dryness, visual acuity (high- and low-contrast), slit-lamp biomicroscopy, posterior lid margin hyperemia, fluorescein tear breakup time, corneal fluorescein staining, conjunctival staining with lissamine green, lid wiper epitheliopathy, meibomian gland expression, keratograph meibography, and Schirmer I test.
  This is a non-randomized, open-label, single-group study evaluating the efficacy and safety of Vevye® for the treatment of clinically significant meibomian gland dysfunction
  Interventions: Drug: Vevye(Cyclosporine 0.1% Ophthalmic Solution)

INTERVENTIONS:
Drug: Vevye(Cyclosporine 0.1% Ophthalmic Solution) — Participants will administer Vevye® (cyclosporine 0.1% ophthalmic solution) twice daily in both eyes for 24 weeks following a 2-week run-in period using a commercially available artificial tear.
  Vevye® contains cyclosporine, a calcineurin inhibitor that reduces ocular surface inflammation, dissolved in a semifluorinated alkane vehicle (perfluorobutylpentane, F4H5), which is preservative-free, water-free, and has no associated pH or osmolarity. The formulation is designed to enhance tear stability and reduce inflammatory processes associated with meibomian gland dysfunction (MGD).
  All participants receive the same treatment in this non-randomized, open-label, single-group interventional trial evaluating the efficacy and safety of Vevye® for MGD.
  Other Names: Vevye®; Cyclopsorine Ophthalmic Solution 0.1%

SUMMARY:
This research study evaluates a prescription eye drop called Vevye® (cyclosporine 0.1%) for adults who have meibomian gland dysfunction (MGD), a common eye condition that can cause dry, irritated, or burning eyes.

If you join the study, after a short "run-in" period using artificial tears, you will receive Vevye twice a day for about 24 weeks (approximately six months). During that time you will attend several clinic visits where your eye symptoms, lid health, tear film, and meibomian gland function will be assessed. The goal is to learn whether Vevye improves symptoms (like eye dryness or irritation) and signs (such as changes on the eye's surface or lid margins) of MGD.

You will also be monitored for safety and comfort of the eye drop. The information obtained from this study may help determine whether this treatment is beneficial for people with this condition and contribute to future care options. Participation is voluntary and you may stop at any time.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, interventional clinical trial designed to evaluate the efficacy of Vevye® (cyclosporine 0.1% ophthalmic solution) for the treatment of clinically significant meibomian gland dysfunction (MGD).

The study begins with a two-week run-in period during which participants use a commercially available artificial tear, followed by a 24-week intervention phase with Vevye® dosed twice daily in both eyes. Clinical examinations occur at screening (Day -14), baseline (Day 0), and at Days 28, 84, and 168.

Approximately 48 adults (age ≥ 18 years) with clinically significant MGD will be enrolled at the University of Alabama at Birmingham, School of Optometry. Each participant will complete five study visits over about six months, lasting approximately 50 to 90 minutes each.

At each visit, standardized ocular assessments are performed, including:

Visual Analog Scale (VAS) Dryness survey,

Habitual visual acuity under high- and low-contrast conditions,

Slit-lamp biomicroscopy and evaluation of posterior lid margin hyperemia,

Fluorescein tear breakup time, corneal fluorescein staining, and conjunctival staining with lissamine green,

Lid wiper epitheliopathy evaluation,

Meibomian gland expression using the Meibomian Gland Evaluator,

Infrared keratograph meibography, and

Schirmer I test without anesthesia.

Primary endpoints include change from baseline to Week 24 in VAS dryness, corneal fluorescein staining (NEI scale), and meibomian gland expressibility. Exploratory endpoints include posterior lid margin hyperemia, lid wiper epitheliopathy, contrast sensitivity, low-contrast visual acuity, fluorescein tear breakup time, conjunctival staining, and gland dropout by meibography.

Participants are trained on dosing technique and use of a dosing diary. Product accountability and log review occur at every visit to monitor compliance. Adverse events are recorded throughout the study, and early termination may occur if clinically indicated.

The most common expected side effects are mild, transient burning, stinging, redness, or blurred vision after instillation. Participants are instructed not to use Vevye® while wearing contact lenses.

There are no direct benefits guaranteed from participation, although some individuals may experience improvement in eye comfort or tear quality. The findings may help determine whether Vevye® is effective for people with MGD and contribute to developing better treatment options for this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. VAS Dryness > 70
3. Posterior lid margin hyperemia grade 2 or worse for both eyes
4. Corneal fluorescein staining > 6 (NEI scale) for at least one eye
5. Modified meibomian gland expression score ≥ 23 for both eyes OR ≥ 7 for expressible glands for both eyes OR a combination of the two
6. Unanesthetized Schirmer ≥ 5 mm in 5 minutes for both eyes

Exclusion Criteria:

1. Age > 18 years
2. VAS Dryness > 70
3. Posterior lid margin hyperemia grade 2 or worse for both eyes
4. Corneal fluorescein staining > 6 (NEI scale) for at least one eye
5. Modified meibomian gland expression score ≥ 23 for both eyes OR ≥ 7 for expressible glands for both eyes OR a combination of the two
6. Unanesthetized Schirmer ≥ 5 mm in 5 minutes for both eyes

4.2 EXCLUSION CRITERIA

1. Contact lens wear within two weeks of study enrollment or planned during study period
2. Habitual visual acuity worse than 0.30 logMAR in either eye
3. Previous or current diagnosis of any of the following conditions:

   1. Sjögren's disease
   2. Stevens-Johnson syndrome
   3. Keratoconus
   4. Herpetic keratitis
   5. Pterygium
   6. Any other condition that in the opinion of the clinician would interfere with study parameters
4. Use of any of the following medications within 30 days of enrollment:

   1. Topical ophthalmic cyclosporine (including but not limited to Restasis®, Cequa®, Vevye®, generic, or compounded versions)
   2. Xiidra®
   3. Miebo®
   4. Tyrvaya
   5. Tryptyr®
   6. Topical ocular steroids
   7. Any topical anti-glaucoma medication
5. Any of the following procedural treatments for MGD within 6 months of enrollment:

   1. LipiFlow®
   2. TearCare®
   3. iLux®
   4. Intense pulsed light (IPL)
   5. Therapeutic gland expression
   6. Any other procedure targeting the meibomian glands
6. Insertion or removal of permanent punctal plugs within 3 months of enrollment
7. Insertion of dissolvable punctal plugs within 9 months of enrollment (or within 3 months of expected dissolution date, if known)
8. Presence of active ocular allergies
9. Previous intraocular surgery within 6 months of enrollment
10. Previous refractive surgery within 2 years of enrollment
11. Current or planned pregnancy during the study period
12. Current or planned lactation during the study period
13. Females of childbearing potential who are not using effective contraception
14. Known allergy or sensitivity to the study drug
15. Dose modification of oral antihistamines or antidepressants within 1 month of enrollment
16. Current enrollment or enrollment within 60 days in any other study of an investigational drug or device
17. Clinical opinion of the study doctor based on clinical examination and/or participant compliance with protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Meibomian Gland Expressibility Score | Baseline to Week 24 (±1 week)
  Meibomian gland function will be quantified using a standardized Meibomian Gland Evaluator. Expressibility is graded based on the quality and quantity of expressed meibum from five glands in each lid region. The change in mean expressibility score from baseline to Week 24 will determine improvement in gland function with Vevye® therapy.
Change in Visual Analog Scale (VAS) Dryness Score | Baseline to Week 24 (±1 week)
  The VAS Dryness assessment measures both the frequency ("rarely" to "all the time") and severity ("very mild" to "very severe") of eye dryness symptoms using 0-100 point horizontal sliders. Each participant's change from baseline to Week 24 will be analyzed to evaluate improvement in subjective dryness associated with meibomian gland dysfunction (MGD).
Change in Corneal Fluorescein Staining (NEI Scale) | Baseline to Week 24 (±1 week)
  Corneal fluorescein staining evaluates epithelial integrity of the cornea using the NEI/Industry scale. Five corneal zones are graded (0-3 each; total 0-15 per eye). The mean change in total corneal fluorescein staining score from baseline to Week 24 will assess ocular surface improvement following Vevye® treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian F Ziemanski, OD, PhD, Principal Investigator — The University of Alabama at Birmingham, School of Optometry
Locations (1):
- University of Alabama at Birmingham, School of Optometry, Clinical Eye Research Facility, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside of the study team, sponsor, or regulatory agencies.
  Participant data will be used only for analysis related to this study and may be reviewed by authorized representatives of the sponsor (Harrow, Inc.), the University of Alabama at Birmingham Institutional Review Board (IRB), and regulatory authorities as required by law.
  De-identified summary results may be shared in aggregate form in publications or presentations, but no individual-level data will be made publicly available.